CLINICAL TRIAL: NCT05588089
Title: The Effect of Baby Care Training Given to Fathers After Birth on Paternal Attachment, Maternal Postpartum Depression and Quality of Life
Brief Title: The Effect of Baby Care Training Given to Fathers After Birth
Acronym: Babycare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Fatma Yildirim, Principal Investigator, Hitit University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: Hitituniversity
Record Dates: First submitted 2022-10-12; First posted 2022-10-20 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Mothers; Fathers
MeSH Terms: interventions — Sensitivity Training Groups

STUDY DESIGN:
Intervention Model Description: The study is of a semi-separate type and all women can be trained.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): After the birth of the control group, the "Personal Information Form for Fathers" and "Infant Care Questionnaire" were applied to the fathers as pre-tests in the clinic. After the training, the fathers will be called at the 2nd, 3rd, 4th, 8th and 12th weeks, and the "Fathers' Participation in Baby Care Chart" will be applied 5 times during 12 weeks. In addition, "Father-Infant Attachment Scale" and "Infant Care Questionnaire" were applied to fathers at 12 weeks as posttests.
  "Personal Information Form for Mothers" will be filled by mothers in the postpartum clinic, mothers are called at 4th, 8th and 12th weeks and "Edinburgh Postpartum Depression Scale" and "Postpartum Quality of Life Scale" are applied.
- Intervention group (Experimental): For the experimental group, "Personal Information Form for Fathers" and "Infant Care Questionnaire" were applied to the fathers in the clinic after birth as a pre-test. In the clinic, baby care training was given to fathers practically in 30-35 minutes. After the applied training, the "Baby Care Training Program Content" prepared by the researchers was given to the fathers. After the training, the fathers were called at the 2nd, 3rd, 4th, 8th and 12th weeks, and the "Paternals' Participation in Baby Care Chart" was applied 5 times during 12 weeks. In addition, the fathers were called at the 12th week and the "Infant Care Questionnaire Form" was applied as a post-test and the "Father-Infant Attachment Scale" was applied.
  "Personal Information Form for Mothers" was applied to the mothers after the birth in the clinic, and the mothers were called at the 4th, 8th and 12th weeks and the "Edinburgh Postpartum Depression Scale" and the "Postpartum Quality of Life Scale" were applied.
  Interventions: Other: Training group

INTERVENTIONS:
Other: Training group — For the experimental group, "Personal Information Form for Fathers" and "Infant Care Questionnaire" were applied to the fathers in the clinic after birth as a pre-test. In the clinic, baby care training was given to fathers practically in 30-35 minutes. After the applied training, the "Baby Care Training Program Content" prepared by the researchers was given to the fathers.
  Arms: Intervention group

SUMMARY:
The aim of this study is to provide infant care training to fathers and to measure father-infant attachment and maternal postpartum depression and quality of life.

DETAILED DESCRIPTION:
Objective: The aim of this study is to provide infant care training to fathers and to measure father-infant attachment and maternal postpartum depression and quality of life.

Design: The data for the study were collected using the introductory information form (IIF) and the father-infant attachment scale (FIAS) for fathers, Edinburgh Postpartum Depression Scale and Postpartum Quality of Life Scale for mothers.

Participants and setting: A total of 64 fathers and 64 mothers, including 32 in the intervention group and 32in the control group who met the inclusion criteria of the study were included randomly.

ELIGIBILITY:
Inclusion Criteria:

* The mother and father are over 18 years old,
* Parents becoming parents for the first time,
* The newborn is healthy, born at term, with the mother and father,
* Parents' knowledge of Turkish,
* Mothers who accepted to participate in the study and received baby care training by participating in the pregnant class,
* Parents' willingness to participate in the research.

Exclusion Criteria:

* Having a baby born as a result of a risky pregnancy,
* The newborn is in intensive care,
* Presence of diagnosed psychiatric disease in the mother and father.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postpartum Depression Scale | 5 months
  The scale is a 4-point Likert type and consists of 10 questions. Each question consists of four options and is scored between 0-3. The lowest score that can be obtained from the scale was reported as 0 and the highest score as 30.

SECONDARY OUTCOMES:
Postpartum Quality of Life Scale | 5 months
  This 6-point Likert type scale; kinship-family-friend, health, psychological, socioeconomic and spouse subscale consists of a total of 5 subscales and a total of 40 items.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Yıldırım, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim F, Sahin E. Does father involvement affect attachment and maternal depression and quality of life?: a randomized controlled trial. Fam Pract. 2025 Apr 12;42(3):cmaf024. doi: 10.1093/fampra/cmaf024. PMID 40317211